CLINICAL TRIAL: NCT06894615
Title: Safety and Efficacy of the BTL-995-rTMS Device for the Reduction of Binge-eating
Brief Title: EXOMIND (BTL-995) for the Reduction of Binge-eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-995_CTCZ100
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-03

CONDITIONS: Binge Eating; Binge-Eating Disorder
Keywords: binge eating; Binge-Eating Disorder; weight loss; ExoTMS; EXOMIND
MeSH Terms: conditions — Bulimia; Binge-Eating Disorder; Weight Loss | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with BTL-995-rTMS (Experimental): Transcranial magnetic stimulation treatment with the BTL-995-rTMS device
  Interventions: Device: Treatment with BTL-995-rTMS

INTERVENTIONS:
Device: Treatment with BTL-995-rTMS — Six transcranial magnetic stimulation treatments with the BTL-995-rTMS device will be delivered over the left dorsolateral prefrontal cortex, spaced 2 to 4 days apart. The intensity will be adjusted according to the subject's feedback, up to 70% of the individual's motor threshold.
  Other Names: EXOMIND (BTL-995) with ExoTMS

SUMMARY:
The goal of this clinical trial is to evaluate if the treatment with the BTL-995-rTMS device is able to reduce binge eating in adults above the age of 22 years. The main question it aims to answer is:

Whether the treatment with the BTL-995-rTMS device reduces binge eating.

Participants will be asked to:

* Undergo six treatments
* Undergo weight measurements
* Complete the Binge Eating Scale
* Complete the Therapy Comfort Questionnaire
* Complete the Satisfaction Questionnaire

DETAILED DESCRIPTION:
This study uses a single-center, single-arm, open-label, interventional design.

Subjects scoring more than 17 points on the Binge Eating Scale will be enrolled and assigned into one experimental study arm. All participants will receive six treatments with the BTL-995-rTMS device, administered 2 to 4 days apart.

Therapy parameters will be adjusted based on patient feedback and comfort, up to 70% of the individual's motor threshold.

Examination for possible adverse effects will be assessed at each visit.

The Binge Eating Scale will be administered before the first treatment, after the last treatment, and at the 1-month follow-up visit after the final session.

The Therapy Comfort Questionnaire will be administered after the last treatment, while the Satisfaction Questionnaire will be given after the last treatment and at the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Scoring more than 17 points based on the BES
* Age > 22 years
* Voluntarily signed informed consent
* Ability to determine the motor threshold of the participant. The participant's motor threshold could be established as the minimum stimulus required to induce contraction of the right thumb
* Subjects willing and able to abstain from partaking in any other weight management treatments other than the study procedure during study participation
* Willingness to comply with study instructions and to return to the clinic for the required visits
* Women of child-bearing potential* are required to use birth control measures during the whole duration of the study

Exclusion Criteria:

* Electronic implants (Implanted stimulator devices in or near the head - rTMS devices are contraindicated for use in patients who have active or inactive implants (including device leads), deep brain stimulators, cochlear implants, ocular implant, and vagus nerve stimulators, implanted devices such as cardiac pacemakers, defibrillators, neurostimulators. Contraindicated use could result in serious injury or death.
* Metallic or other magnetic sensitive implants/objects in or near the head - rTMS devices are contraindicated for use in patients who have conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head or within 30 cm of the treatment coil. (Examples include implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewellery and hair barrettes. Failure to follow this restriction could result in serious injury or death.)
* Drug pump(s)
* Persons with a tendency to seizure (hypotonic, epileptic)
* Ongoing anticoagulation therapy
* Ongoing severe or life-threatening condition
* Pulmonary insufficiency
* Heart disorders
* Renal insufficiency
* Decompensated hemorrhagic conditions, blood coagulation disorders, cardiovascular diseases
* Malignant or benign tumour
* Fever
* Facial tattoos with metallic ink (within 30 cm of the treatment coil)
* Pregnancy or nursing
* Ongoing intake disorders such as bulimia or anorexia, borderline personality disorder, major depression (elevated seizure risk) or bipolar disorder Personal history of epilepsy
* Personal history of syncope (except the reflex syncope)
* Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without a history of seizure, and without anticonvulsant medication
* Withdrawal from one of the following drugs could form a relative hazard for the application of rTMS due to the resulting significant seizure threshold lowering potential: (e.g. alcohol, barbiturates, benzodiazepines, meprobamate, chloralhydrate etc.)
* Systemic infection
* Patients with a broad range of neuropsychiatric diseases are at elevated risk for seizures. Essentially all neurologic conditions with structural cerebral damage (e.g. stroke, multiple sclerosis, traumatic brain injury, Alzheimer's and other neurodegenerative diseases, meningoencephalitis or intracerebral abscess, parenchymal or leptomeningeal cancers) are associated with an elevated risk for seizures
* History of hyponatremia, hypocalcemia, hypomagnesemia, hypoglycemia, hyperglycemia, renal failure/uremia, liver failure
* History of tendency for raised blood concentrations of pro-convulsant medications due to reduced clearance (e.g. secondary to initiation of antibiotics for treatment of infections)
* Immunosuppressive therapy with cyclosporine, tacrolimus and other agents that can cause the posterior reversible leukoencephalopathy syndrome
* The use of amphetamines, barbiturates, cocaine metabolites, opiates and phencyclidine 72 hours before the therapy.
* Contradictions for the testing used in the trial, for example, the motor threshold cannot be found or quantified.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Change in Binge Eating | 15 months
  The change in the score obtained from the Binge Eating Scale will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, and at the1-month follow-up visit. The score ranges from 0 to 46 and higher scores indicate more frequent and severe binge eating. An improvement is defined as a decrease in score.

SECONDARY OUTCOMES:
Assessment of Therapy Comfort | 15 months
  Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. The Therapy Comfort questionnaire will be administered after the last treatment. Therapy Comfort questionnaire consists of the question "I found the treatment comfortable", to which responses are based on a 5-point Likert scale (1 = "strongly disagree", and 5 = "strongly agree") and the 10-point Numeric Analog Scale for pain (0 = no pain, 10 = worst possible pain"). A higher score for the statement "I found the treatment comfortable", and lower score on the Numeric Analog Scale for pain indicate higher therapy comfort.
Assessment of Satisfaction | 15 months
  Subject Satisfaction with treatment outcomes will be assessed using 5-point Likert Scale Satisfaction questionnaire. The questionnaire will be administered after the last treatment, and at the 1-month follow-up visits. Responses to questions about binge eating and satisfaction with the treatment outcomes will range from "strongly agree" (5 points) to "strongly disagree" (1 point). A higher score for each statement indicate better outcomes.
Incidence of Treatment-related Adverse Events | 15 months
  Monitoring of adverse reactions and side effects will be performed for the evaluation of safety of the treatment with the BTL-995-rTMS device for the reduction of binge eating and to identify side effects and adverse events associated with the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- DP Neuro s.r.o., Prague, Czechia